CLINICAL TRIAL: NCT07203755
Title: A Randomized, Partially Blinded, Dose-Exploratory, Active/Placebo-Controlled Phase I Clinical Trial Evaluating the Safety and Immunogenicity of the Adsorbed Acellular Pertussis (Tricomponent) DPT-Hib (Conjugate)-ACYW135-Group B Meningococcal (Conjugate) Combined Vaccine in Individuals Aged 2 Months to 6 Years
Brief Title: Clinical Trial of the Adsorbed Acellular Pertussis (Tricomponent) DTaP-Haemophilus Influenzae Type b (Conjugate)-ACYW135 Group Meningococcal (Conjugate) Combined Vaccine
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: CanSino Biologics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CTP-DHMCV-001
Record Dates: First submitted 2025-09-25; First posted 2025-10-02 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-09

CONDITIONS: Diphtheria, Tetanus and Acellular Pertussis; Epidemic Meningitis; Haemophilus Influenzae Type B Infection
Keywords: Combined Vaccine; Safety; Immunogenicity; Ages 2 months to 6 years
MeSH Terms: conditions — Diphtheria; Tetanus; Meningitis, Meningococcal; Haemophilus Infections | interventions — Vaccines, Combined; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Part One: Partial Blind Method Design Part Two: Blind Method Design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (11):
- Part I, 1A, low dose, 6 year-old (Experimental): One dose of DTcP-Hib-MCV4 on Day 0
  Interventions: Biological: Adsorbed Acellular Pertussis (3-Component) Diphtheria-Tetanus-Pertussis-Haemophilus influenzae type b (Conjugate)-Meningococcal Group ACYW135 (Conjugate) Combined Vaccine (DTcP-Hib-MCV4)
- Part I, 2A, low dose, 18~24 month-old (Experimental): One dose of DTcP-Hib-MCV4 on Day 0
  Interventions: Biological: DTcP-Hib-MCV4
- Part I, 2B, high dose, 18~24 month-old (Experimental): One dose of DTcP-Hib-MCV4 on Day 0
  Interventions: Biological: DTcP-Hib-MCV4
- Part I, 3A, low dose, 2 month-old (Experimental): 3 doses of DTcP-Hib-MCV4 at 0, 2, and 4 months, followed by a booster dose at 18-24 months of age.
  Interventions: Biological: DTcP-Hib-MCV4
- Part I, 3B, high dose, 2 month-old (Experimental): 3 doses of DTcP-Hib-MCV4 at 0, 2, and 4 months, followed by a booster dose at 18-24 months of age.
  Interventions: Biological: DTcP-Hib-MCV4
- Part I, 3C, 2 month-old (Active Comparator): 3 doses of DTcP at 0, 2, and 4 months, followed by a booster dose at 18-24 months of age.
  Interventions: Biological: Adsorbed Acellular Pertussis (3-Component) Diphtheria-Tetanus-Pertussis (DTcP)
- Part I, 3D, 2 month-old (Active Comparator): 3 doses of Hib at 0, 2, and 4 months, followed by a booster dose at 18-24 months of age.
  Interventions: Biological: Haemophilus influenzae type b (Conjugate) (Hib)
- Part I, 3E, 2 month-old (Active Comparator): 3 doses of MCV4 at 0, 2, and 4 months, followed by a booster dose at 18-24 months of age.
  Interventions: Biological: Meningococcal Group ACYW135 (Conjugate) (MCV4)
- Part I, 4A, 3 month-old (Active Comparator): 3 doses of MCV4 at 0, 1, and 2 months, followed by a booster dose at 12 months of age.
  Interventions: Biological: MCV4
- Part II, Vaccine Group, 2 month-old (Experimental): 3 doses of MCV4 at 0, 2, and 4 months.
  Interventions: Biological: MCV4
- Part II, Placebo Group, 2 month-old (Placebo Comparator): 3 doses of NS at 0, 2, and 4 months.
  Interventions: Other: Sodium Chloride Injection (0.9%) (Saline Solution) (NS)

INTERVENTIONS:
Biological: Adsorbed Acellular Pertussis (3-Component) Diphtheria-Tetanus-Pertussis-Haemophilus influenzae type b (Conjugate)-Meningococcal Group ACYW135 (Conjugate) Combined Vaccine (DTcP-Hib-MCV4) — 1 dose of DTcP-Hib-MCV4 vaccine (0.5ml) on day 0
  Arms: Part I, 1A, low dose, 6 year-old
Biological: DTcP-Hib-MCV4 — 1 dose of DTcP-Hib-MCV4 vaccine (0.5ml) on day 0
  Arms: Part I, 2A, low dose, 18~24 month-old
Biological: DTcP-Hib-MCV4 — 1 dose of DTcP-Hib-MCV4 vaccine (0.5ml) on day 0
  Arms: Part I, 2B, high dose, 18~24 month-old
Biological: DTcP-Hib-MCV4 — 3 doses of DTcP-Hib-MCV4 (0.5ml) at 0, 2, and 4 months, followed by a booster dose at 18-24 months of age.
  Arms: Part I, 3A, low dose, 2 month-old
Biological: DTcP-Hib-MCV4 — 3 doses of DTcP-Hib-MCV4 (0.5ml) at 0, 2, and 4 months, followed by a booster dose at 18-24 months of age.
  Arms: Part I, 3B, high dose, 2 month-old
Biological: Adsorbed Acellular Pertussis (3-Component) Diphtheria-Tetanus-Pertussis (DTcP) — 3 doses of DTcP (0.5ml) at 0, 2, and 4 months, followed by a booster dose at 18-24 months of age.
  Arms: Part I, 3C, 2 month-old
Biological: Haemophilus influenzae type b (Conjugate) (Hib) — 3 doses of Hib (0.5ml) at 0, 2, and 4 months, followed by a booster dose at 18-24 months of age.
  Arms: Part I, 3D, 2 month-old
Biological: Meningococcal Group ACYW135 (Conjugate) (MCV4) — 3 doses of MCV4 (0.5ml) at 0, 2, and 4 months, followed by a booster dose at 18-24 months of age.
  Arms: Part I, 3E, 2 month-old
Biological: MCV4 — 3 doses of MCV4 (0.5ml) at 0, 1, and 2 months, followed by a booster dose at 12 months of age.
  Arms: Part I, 4A, 3 month-old
Biological: MCV4 — 3 doses of MCV4 (0.5ml) at 0, 2, and 4 months.
  Arms: Part II, Vaccine Group, 2 month-old
Other: Sodium Chloride Injection (0.9%) (Saline Solution) (NS) — 3 doses of NS (0.5ml) at 0, 2, and 4 months.
  Arms: Part II, Placebo Group, 2 month-old

SUMMARY:
This clinical trial is conducted in two parts. Part One employs a randomized, partially blinded, dose-escalation, partially active-controlled design. Part Two utilizes a randomized, blinded, placebo-controlled design. Part One is divided into four stages based on age and vaccine dose levels. Part Two consists of the 2-month-old vaccine/placebo groups.

ELIGIBILITY:
Inclusion Criteria:

General Inclusion Criteria:

* Participants aged 2 months (60-89 days), 3 months (90-119 days), 18-24 months, and 6 years of age, with legal guardians or authorized representatives willing to provide identification documentation;
* Legal guardians or authorized representatives provide informed consent, voluntarily sign the informed consent form, and are able to comply with the requirements of the clinical trial protocol;

Part I: Specific Inclusion Criteria:

* Individuals aged 18-24 months who have completed a 3-dose DTaP-containing vaccine series and a meningococcal-containing vaccine primary series, but have not received a DTaP-containing booster dose;
* Individuals aged 6 years who have completed 4 doses of DTaP-containing vaccine but have not received the 5th DTaP-containing vaccine dose; and have only completed the first meningococcal-containing vaccine booster dose, without receiving the second meningococcal-containing vaccine booster dose at age 6.

Exclusion Criteria:

General Exclusion Criteria for First Dose：

* Infants born prematurely (delivery before 37 weeks gestation) or with low birth weight (<2500g) at 2 months (60-89 days) or 3 months (90-119 days) of age;
* Infants aged 2 months (60-89 days) or 3 months (90-119 days) with history of abnormal labor, asphyxia requiring resuscitation, or neurological impairment;
* Severe congenital malformations or developmental disorders, genetic defects, or severe malnutrition;
* History of severe adverse reactions or anaphylaxis to vaccines or vaccine components, such as urticaria, dyspnea, angioedema;
* History of epilepsy, convulsions, seizures, cerebral palsy, psychiatric disorders, or family history thereof; or history of progressive neurological diseases (e.g., Guillain-Barré syndrome, brachial plexus neuritis);
* Diagnosed with congenital or acquired immunodeficiency, HIV infection, lymphoma, leukemia, systemic lupus erythematosus (SLE), juvenile rheumatoid arthritis (JRA), or other autoimmune diseases;
* Acute illness (e.g., fever ≥38.5°C, diarrhea) or acute exacerbation of chronic disease within 3 days prior to receiving the investigational product;
* Known or suspected severe chronic diseases (including: severe respiratory disease, severe cardiovascular disease, liver/kidney disease, severe dermatology conditions, malignancies, etc.);
* Current anal abscess or severe eczema;
* Clinically diagnosed coagulation disorders (e.g., factor deficiency, bleeding disorders, platelet abnormalities) or significant bruising/coagulation impairment;
* Asplenia, functional asplenia, or splenectomy due to any cause;
* Continuous treatment with immunosuppressants, immunomodulators, or cytotoxic agents (exceeding 10 days) within the past 6 months; inhaled or topical steroids are permitted;
* Receipt of blood products or immunoglobulins (excluding hepatitis B immunoglobulin) within the past 3 months;
* Received an injectable live attenuated vaccine within 14 days, or any other vaccine within 7 days;
* Taken antipyretic analgesics or antiallergic medications within 3 days;
* Fever present prior to vaccination, with axillary temperature ≥37.3°C (99.3°F);
* Plans to participate in or is currently participating in any other drug/vaccine clinical trial;
* Any other factors deemed by the investigator to make the subject unsuitable for participation in the clinical trial.

Part I: Exclusion Criteria for the First Dose：

* Infants aged 2 months (60-89 days) who have received vaccines containing meningococcal, DTP, or Haemophilus influenzae type b components;
* Infants aged 3 months (90-119 days) who have received a vaccine containing meningococcal components;
* Individuals aged 18-24 months who have received vaccines containing meningococcal or Haemophilus influenzae type b components within the past six months;
* Individuals aged 18-24 months with abnormal pre-vaccination blood count or urinalysis results deemed clinically significant by the investigator;
* Children aged 6 years who, prior to vaccination, exhibit abnormal results in relevant indicators of complete blood count, blood biochemistry, coagulation function, or urinalysis, and are deemed clinically significant by the investigator;
* Individuals with a history of any of the following diseases: meningococcal meningitis, Haemophilus influenzae type b disease, pertussis, diphtheria, or tetanus.

Part II: Specific Exclusion Criteria for the First Dose

* History of vaccination with any meningococcal-containing vaccine;
* History of meningococcal disease. General Exclusion Criteria for Subsequent Doses：
* Occurrence of a serious adverse event related to vaccination following the previous dose;
* Vaccine-related Grade 3 or higher allergic reaction following the previous dose;
* Any other factors deemed by the investigator to make the subject unsuitable for continued participation in the clinical trial.

Ages: 2 Months to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 260 (Estimated)
Dates: Start 2025-12-19 (Actual); Primary Completion 2029-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse reactions | Parts I and II: Within 14 days after each dose

SECONDARY OUTCOMES:
Incidence of adverse events | Part I Sections 1A, 2A, 2B: Within 14 days after exemption
Incidence of adverse events | Part I Sections 3A, 3B, 3C, 3D, 3E, 4A and Part II: Within 14 days after each dose
Incidence of adverse reactions/events | Part I Sections 1A, 2A, 2B: Within 30 minutes after exemption
Incidence of adverse reactions/events | Part I Sections 3A, 3B, 3C, 3D, 3E, 4A and Part II: Within 30 minutes after each dose
Incidence of adverse reactions/events | Part I Sections 1A, 2A, 2B: Within 30 days after exemption
Incidence of adverse reactions/events | Part I Sections 3A, 3B, 3C, 3D, 3E, 4A and Part II: Within 30 days after each dose
Incidence of Serious Adverse Event (SAE) | Part I Sections 1A, 2A, 2B: Within 180 days after exemption
Incidence of Adverse Event of Special Interest (AESI) | Part I Sections 1A, 2A, 2B: Within 180 days after exemption
Incidence of Serious Adverse Event (SAE) | Part I Sections 3A, 3B, 3C, 3D, 3E, 4A and Part II: Within 180 days after the first dose to the booster dose
Incidence of Adverse Event of Special Interest (AESI) | Part I Sections 3A, 3B, 3C, 3D, 3E, 4A and Part II: Within 180 days after the first dose to the booster dose
Abnormal laboratory test values | Part I Sections 1A, 2A, 2B: 4 days after exemption
Seroconversion Rate of A, C, Y, W135 Group Meningococcal Antibody | Part I Sections 3A, 3B, 3C, 3D, 3E, 4A: 30 days after primary vaccination, 30 days before and after booster vaccination
Geometric Mean Titer (GMT) of A, C, Y, W135 Group Meningococcal Antibody | Part I Sections 3A, 3B, 3C, 3D, 3E, 4A: 30 days after primary vaccination, 30 days before and after booster vaccination, at the age 3
Positive Rate of A, C, Y, W135 Group Meningococcal Antibody | Part I Sections 3A, 3B, 3C, 3D, 3E, 4A: 30 days after primary vaccination, 30 days before and after booster vaccination, at the age 3
Geometric mean increase (GMI) of A, C, Y, W135 Group Meningococcal Antibody | Part I Sections 3A, 3B, 3C, 3D, 3E, 4A: 30 days after primary vaccination, 30 days before and after booster vaccination, at the age 3
Proportion of individuals with ≥1:128 titers for A, C, Y, W135 Group Meningococcal Antibody | Part I Sections 3A, 3B, 3C, 3D, 3E, 4A: 30 days after primary vaccination, 30 days before and after booster vaccination, at the age 3
Seroconversion rates of serum anti-Pertussis Toxoid (PT), Filamentous hemagglutmin (FHA), Pertactin (PRN), Diphtheria Toxoid (DT), Tetanus Toxoid (TT) antibody | Part I Sections 3A, 3B, 3C, 3D, 3E: 30 days after primary vaccination, 30 days before and after booster vaccination, at the age 3
Geometric Mean Concentration (GMC) of serum anti-PT, FHA, PRN, DT, TT antibody | Part I Sections 3A, 3B, 3C, 3D, 3E: 30 days after primary vaccination, 30 days before and after booster vaccination, at the age 3
Seropositivity rate of serum anti-PT, FHA, PRN, DT, TT antibody | Part I Sections 3A, 3B, 3C, 3D, 3E: 30 days after primary vaccination, 30 days before and after booster vaccination, at the age 3
GMI of serum anti-PT, FHA, PRN, DT, TT antibody | Part I Sections 3A, 3B, 3C, 3D, 3E: 30 days after primary vaccination, 30 days before and after booster vaccination, at the age 3
Percentage of serum anti-Hib-Polyribosyl Ribitol Phosphate (PRP) antibody concentrations ≥0.15 μg/ml | Part I Sections 3A, 3B, 3C, 3D, 3E: 30 days after primary vaccination, 30 days before and after booster vaccination, at the age 3
Percentage of serum anti-Hib-PRP antibody concentrations ≥1.0 μg/ml | Part I Sections 3A, 3B, 3C, 3D, 3E: 30 days after primary vaccination, 30 days before and after booster vaccination, at the age 3
GMC of serum anti-Hib-PRP antibodies | Part I Sections 3A, 3B, 3C, 3D, 3E: 30 days after primary vaccination, 30 days before and after booster vaccination, at the age 3
Seroconversion rate of serum anti-Hib-PRP antibodies | Part I Sections 3A, 3B, 3C, 3D, 3E: 30 days after primary vaccination, 30 days before and after booster vaccination, at the age 3
GMI of serum anti-Hib-PRP antibodies | Part I Sections 3A, 3B, 3C, 3D, 3E: 30 days after primary vaccination, 30 days before and after booster vaccination, at the age 3

CONTACTS AND LOCATIONS:
Overall Officials: Yanxia Wang, Principal Investigator — Henan Center for Disease Control and Prevention
Locations (1):
- Liangyuan District Center for Disease Control and Prevention, Shangqiu City, Shangqiu, Henan, China